CLINICAL TRIAL: NCT02057510
Title: Clinical Registry of Dental Outcomes in Head and Neck Cancer Patients
Brief Title: Observational Study of Dental Outcomes in Head and Neck Cancer Patients
Acronym: ORARAD
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Minnesota (Other); UConn Health (Other); University of Pennsylvania (Other); Brigham and Women's Hospital (Other); NYU Langone Health (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 12-040-E; 1U01DE022939-01 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Dental Disease; Xerostomia; Osteoradionecrosis
Keywords: Head and Neck Cancer; Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatognathic Diseases; Xerostomia; Osteoradionecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients receiving head and neck RT: No intervention

SUMMARY:
The purpose of this study is to measure the two-year rate of tooth loss in patients who have received external beam radiation therapy with curative intent for head and neck cancer. The study will also evaluate the sequelae of radiation therapy and oral complications that may occur as a result to receiving radiation therapy.

DETAILED DESCRIPTION:
This is a prospective cohort study to document dental and other oral outcomes in patients who receive external beam radiation therapy with curative intent, as part of clinical care for a head and neck cancer. Five hundred and seventy-five participants will be enrolled. All study participants will receive a baseline oral examination prior to the start of radiation therapy. Follow-up examinations and data collection will be conducted at six-month intervals up to 2 years after the start of radiation therapy. The primary outcome will be the two-year rate of tooth loss. Secondary outcomes will include measures of dental caries, periodontal health, salivary flow, and exposed bone/osteoradionecrosis.

The proposed research will provide more information to inform the community about the sequelae of Radiation Therapy (RT) in head and neck cancer patients, to refine current guidelines and to design future studies on the dental management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older;
* Willing and able to provide signed and dated consent form;
* Diagnosed with head and neck squamous cell carcinoma (SCC) or a salivary gland cancer (SGC), and intends to receive external beam radiation therapy (RT) with curative intent (tumor eradication), with or without concomitant chemotherapy;

OR

* Diagnosed with a non-SCC, non-SGC malignancy of the head and neck region, and intends to receive RT, with or without concomitant chemotherapy. The subject must be expected to receive at least 4500 cGy to one of the following sites:

  1. base of tongue
  2. buccal/labial mucosa
  3. epiglottis
  4. floor of mouth
  5. gingiva/alveolar ridge
  6. hard palate
  7. hypopharynx
  8. larynx
  9. lip
  10. mandible
  11. maxilla
  12. maxillary sinus
  13. nasal cavity
  14. nasopharynx
  15. neck
  16. oral cavity
  17. oral tongue
  18. oropharynx
  19. paranasal sinus/orbit
  20. parotid gland
  21. pharynx
  22. retromolar trigone
  23. soft palate
  24. sublingual gland
  25. submandibular gland
  26. tonsil;
* At least 1 natural tooth remaining or expected to remain in the mouth after completion of the pre-RT dental extractions, if any;
* Willing to comply with all study procedures;
* Willing to participate for the duration of the study.

Exclusion Criteria:

* Receiving palliative RT;
* History of prior curative RT to the head and neck region to eradicate a malignancy;
* Incarcerated at time of screening;
* Anything that would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and Neck Radiation Oncology patients
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2014-02; Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Tooth loss | Two Years
  The primary outcome measure is the two-year rate of tooth loss in patients who have received at least one session of external beam radiation therapy with curative intent for head and neck cancer.
  "Tooth loss" will be defined as a dental extraction that has been performed or recommended. Since dental extractions are often avoided in this population because of the increased risk of osteoradionecrosis (ORN), tooth loss will also include teeth having a dental procedure to avoid extraction of a tooth that would otherwise have been extracted if the individual had not received RT and teeth recommended for extraction that have not been treated. The following categories will constitute teeth that would otherwise be recommended for extraction:
  * non-restorable because of fracture or extent of caries;
  * amputated crown with root remaining;
  * uncontrolled or persistent periodontal or odontogenic infection.

SECONDARY OUTCOMES:
Incidence of exposed intraoral bone | Two Years
  Two year incidence of exposed intraoral bone, suggestive of ORN. This will be defined as exposed maxillary or mandibular bone with an avascular appearance in a quadrant that has received RT
Extraction complications | Within 14 days following procedure
  Incidence of post-extraction complications
Decayed, Missing or Filled Surfaces (DMFS) Index | Baseline, 24 months
  Two year change in DMFS - Decayed, Missing or Filled Surfaces Index
Periodontal Measures | Baseline, 24 months
  Two year change in periodontal measures
Stimulated Salivary Flow Rate | Baseline, 18 months
  18 month changes in stimulated whole salivary flow rates
Trismus measure | Baseline, 24 months
  Two year change in mouth opening in mm
Topical fluoride use for caries prevention | Baseline, 24 months
  Two year use of fluoride to prevent new caries
Chronic Oral Mucositis Incidence | Baseline, 24 months
  Two year chronic oral mucositis incidence
Quality of Life after Radiation Therapy | Baseline, 24 months
  Two year change in radiation therapy-specific quality of life measures
Oral Cancer Pain Scale | Baseline, 24 months
  Two year change in pain scores as measured with the University of California at San Francisco (UCSF) oral cancer pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Brennan, DDS, MHS, Study Chair — Wake Forest University Health Sciences; Rajesh Lalla, DDS, PhD, Study Chair — University of Connecticut Health Center - School of Dental Medicine
Locations (6):
- United States (6):
  - University of Connecticut Health Center - School of Dental Medicine, Farmington, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New York University - College of Dentistry, New York, New York
  - University of North Carolina - School of Dentistry, Chapel Hill, North Carolina
  - Carolinas Medical Center - Dental Clinic, Charlotte, North Carolina
  - University of Pennsylvania - School of Dental Medicine, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Brennan MT, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Mohammadi K, Long Simpson L, Voelker H, Hodges JS, Lalla RV. Dental disease before radiotherapy in patients with head and neck cancer: Clinical Registry of Dental Outcomes in Head and Neck Cancer Patients. J Am Dent Assoc. 2017 Dec;148(12):868-877. doi: 10.1016/j.adaj.2017.09.011. PMID 29173331
- [Result] Lalla RV, Treister N, Sollecito T, Schmidt B, Patton LL, Mohammadi K, Hodges JS, Brennan MT; OraRad Study Group. Oral complications at 6 months after radiation therapy for head and neck cancer. Oral Dis. 2017 Nov;23(8):1134-1143. doi: 10.1111/odi.12710. Epub 2017 Aug 3. PMID 28675770
- [Result] Lalla RV, Long-Simpson L, Hodges JS, Treister N, Sollecito T, Schmidt B, Patton LL, Brennan MT; OraRad Study Group. Clinical registry of dental outcomes in head and neck cancer patients (OraRad): rationale, methods, and recruitment considerations. BMC Oral Health. 2017 Feb 27;17(1):59. doi: 10.1186/s12903-017-0344-y. PMID 28241807
- [Result] Brennan MT, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Yang Y, Lin A, Elting LS, Hodges JS, Lalla RV. Epidemiologic factors in patients with advanced head and neck cancer treated with radiation therapy. Head Neck. 2021 Jan;43(1):164-172. doi: 10.1002/hed.26468. Epub 2020 Sep 29. PMID 32991009
- [Result] Talevi V, Wen J, Lalla RV, Brennan MT, Mougeot FB, Mougeot JC. Identification of single nucleotide pleomorphisms associated with periodontal disease in head and neck cancer irradiation patients by exome sequencing. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Jul;130(1):32-42.e4. doi: 10.1016/j.oooo.2020.02.013. Epub 2020 May 22. PMID 32451231
- [Result] Mougeot JC, Stevens CB, Almon KG, Paster BJ, Lalla RV, Brennan MT, Mougeot FB. Caries-associated oral microbiome in head and neck cancer radiation patients: a longitudinal study. J Oral Microbiol. 2019 Mar 8;11(1):1586421. doi: 10.1080/20002297.2019.1586421. eCollection 2019. PMID 30891159
- [Result] Brennan MT, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Lin A, Elting LS, Hodges JS, Lalla RV. Tooth Failure Post-Radiotherapy in Head and Neck Cancer: Primary Report of the Clinical Registry of Dental Outcomes in Head and Neck Cancer Patients (OraRad) Study. Int J Radiat Oncol Biol Phys. 2022 Jun 1;113(2):320-330. doi: 10.1016/j.ijrobp.2021.11.021. Epub 2021 Dec 5. PMID 34879248
- [Result] Lalla RV, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Helgeson ES, Lin A, Rybczyk C, Dowsett R, Hegde U, Boyd TS, Duplinsky TG, Brennan MT. Radiation therapy for head and neck cancer leads to gingival recession associated with dental caries. Oral Surg Oral Med Oral Pathol Oral Radiol. 2022 May;133(5):539-546. doi: 10.1016/j.oooo.2022.01.016. Epub 2022 Jan 31. PMID 35304084
- [Result] Brennan MT, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Lin A, Elting LS, Helgeson ES, Lalla RV. Dental Caries Postradiotherapy in Head and Neck Cancer. JDR Clin Trans Res. 2023 Jul;8(3):234-243. doi: 10.1177/23800844221086563. Epub 2022 Apr 11. PMID 35403479
- [Result] Lin A, Helgeson ES, Treister NS, Schmidt BL, Patton LL, Elting LS, Lalla RV, Brennan MT, Sollecito TP. The impact of head and neck radiotherapy on salivary flow and quality of life: Results of the ORARAD study. Oral Oncol. 2022 Apr;127:105783. doi: 10.1016/j.oraloncology.2022.105783. Epub 2022 Feb 26. PMID 35231809
- [Result] Treister NS, Brennan MT, Sollecito TP, Schmidt BL, Patton LL, Mitchell R, Haddad RI, Tishler RB, Lin A, Shadick R, Hodges JS, Lalla RV. Exposed bone in patients with head and neck cancer treated with radiation therapy: An analysis of the Observational Study of Dental Outcomes in Head and Neck Cancer Patients (OraRad). Cancer. 2022 Feb 1;128(3):487-496. doi: 10.1002/cncr.33948. Epub 2021 Oct 19. PMID 34665873
- [Result] Ward MC, Carpenter MD, Noll J, Carrizosa D, Moeller BJ, Helgeson ES, Lalla RV, Brennan MT. Oncologists' Perspective on Dental Care Around the Treatment of Head and Neck Cancer: A Pattern of Practice Survey. JCO Oncol Pract. 2022 Jan;18(1):e28-e35. doi: 10.1200/OP.20.00913. Epub 2021 Jul 9. PMID 34242067
- [Result] Threet EJ, Napenas JJ, Petersen C, Mitchell R, Long-Simpson L, Shadick R, Valentino KC, Rybczyk CA, Blake JA, Brown MC, Aidoo R, Helgeson ES, Lalla RV, Brennan MT. Survey of experiences and barriers to dental care post-head and neck cancer in OraRad study participants. Oral Surg Oral Med Oral Pathol Oral Radiol. 2023 Apr;135(4):501-509. doi: 10.1016/j.oooo.2022.11.011. Epub 2022 Dec 13. PMID 36717342
- [Result] Lalla RV, Hodges JS, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Lin A, Brennan MT. Tooth-level predictors of tooth loss and exposed bone after radiation therapy for head and neck cancer. J Am Dent Assoc. 2023 Jun;154(6):519-528.e4. doi: 10.1016/j.adaj.2023.03.009. PMID 37236706
- [Result] Patton LL, Helgeson ES, Brennan MT, Treister NS, Sollecito TP, Schmidt BL, Lin A, Chera BS, Lalla RV. Oral health-related quality of life after radiation therapy for head and neck cancer: the OraRad study. Support Care Cancer. 2023 Apr 20;31(5):286. doi: 10.1007/s00520-023-07750-2. PMID 37079106